CLINICAL TRIAL: NCT00230698
Title: Topiramate (RWJ-17021-000) Monotherapy Clinical Trial in Patients With Recently Diagnosed Partial-Onset Seizures
Brief Title: A Study of the Effectiveness and Safety of Topiramate Monotherapy in Patients With Recently Diagnosed Partial-Onset Seizure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR002503
Record Dates: First submitted 2005-09-29; First posted 2005-10-03 (Estimated); Last update posted 2010-11-15 (Estimated); Status verified 2010-11

CONDITIONS: Epilepsy; Epilepsies, Partial; Seizures
Keywords: Epilepsy; Partial Epilepsies; Seizures; Topiramate
MeSH Terms: conditions — Epilepsy; Epilepsies, Partial; Seizures | interventions — Topiramate

INTERVENTIONS:
Drug: topiramate

SUMMARY:
The purposes of this study are (1) to compare the effectiveness of two doses of topiramate and (2) to assess the safety of topiramate alone in the treatment of pediatric and adult patients with recently diagnosed epilepsy characterized by partial-onset seizures.

DETAILED DESCRIPTION:
Topiramate is approved for treating epilepsy in combination with other epilepsy drugs, but not approved for treating epilepsy as sole treatment or in recently diagnosed epilepsy characterized by partial-onset seizures. This is a randomized, double-blind, parallel-group, multicenter trial to investigate the effectiveness and safety of topiramate in pediatric and adult patients with recently diagnosed epilepsy characterized by partial-onset seizures. There are four phases of this trial: Retrospective Baseline, Open-Treatment, Double-Blind, and Long-Term Extension. During the Retrospective Baseline Phase, eligibilities of the potential patients are evaluated. During the Open-Treatment Phase, patients receive 25 milligrams[mg] daily of topiramate to assess their ability to tolerate the medication. During the Double-Blind Phase, patients are randomized to a high or a low dose of topiramate. Patients continue to receive the study medication until one of the following occurs: (1) treatment fails; (2) 4 months have passed since the last patient was randomized; or (3) the patient withdraws from the study. Unless withdrawn from the study, the patient may enter the Long-Term Extension Phase and receive high dose topiramate (maximum of either 1,600mg daily for patients >= 14 years of age, or 24mg/kilogram[kg] for patients < 14 years of age) until the patient withdraws or the study is stopped by the sponsor. The study hypothesis is that topiramate will be effective and well tolerated in treating pediatric and adult patients with recently diagnosed epilepsy characterized by partial-onset seizures. Open-Treatment: topiramate 25mg daily by mouth for 7days. Double-Blind: low dose (50 mg or 25mg daily, depending on body weight) or high dose (500mg or 200mg daily, depending on body weight) for up to 4 months. Long-Term Extension: high dose (1600mg or 24mg/kg daily, maximum) for various duration.

ELIGIBILITY:
Inclusion Criteria:

* Body weight between 25 kg and 110 kg (approximately 55-240 lb)
* Diagnosis of epilepsy characterized by unprovoked partial-onset seizures that were diagnosed within the past three years
* During the three-month Retrospective Baseline Phase, patients must have had at least one seizure, have had an average of no more than two seizures per month, and have had no more than three seizures in any given month. None of the seizures should occur in a cluster pattern
* During the three-month Retrospective Baseline Phase, patients must receive either no other standard Anti-Epileptic Drug (AED), or be on one AED
* Patients currently on one AED must be considered inadequately controlled
* Must have evidence from computed tomography (CT) or magnetic resonance imaging (MRI) of the absence of an arteriovenous malformation or a progressive lesion such as a tumor.

Exclusion Criteria:

* Patients who do not have epilepsy, such as patients with pseudoseizures or a treatable cause of seizures
* Patients with benign rolandic epilepsy
* Patients with progressive or degenerative disorders
* Patients with a documented history of generalized tonic-clonic status epilepticus during the three month Retrospective Baseline Phase
* Patients with a significant history (within the past two years) of medical disease that may impair their reliable participation in the trial or necessitate the use of medication not allowed by this protocol
* Patients who are unable to take their medication either independently or with assistance.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 1995-11; Study Completion 2002-08 (Actual)

PRIMARY OUTCOMES:
Time to exit during the double blind phase (2 partial onset seizures with or without a secondarily generalized component, a secondarily generalized tonic clonic seizure when none existed prior to this phase, or 1 episode of status epilepticus).

SECONDARY OUTCOMES:
Laboratory, vital signs, electrocardiogram data and adverse events reported during the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Gilliam FG, Veloso F, Bomhof MA, Gazda SK, Biton V, Ter Bruggen JP, Neto W, Bailey C, Pledger G, Wu SC. A dose-comparison trial of topiramate as monotherapy in recently diagnosed partial epilepsy. Neurology. 2003 Jan 28;60(2):196-202. doi: 10.1212/01.wnl.0000048200.12663.bc. PMID 12552030